CLINICAL TRIAL: NCT04594096
Title: Improving Treatment-Related Symptom Management in Adolescents and Young Adults
Brief Title: Improving Treatment-Related Symptom Management in Adolescents and Young Adults With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1575166
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: 2 telehealth visits with a medical provider (either an MD or NP) after last chemotherapy administration in the cycle, or as otherwise indicated
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Arm (Experimental): Observation periods will be from 4 days post last administration of chemotherapy until the next chemotherapy administration.
  All patients will undergo an initial observation period that will span two chemotherapy cycles and will be receiving clinical care as usual determined by the primary oncology team.
  Patients enrolled on the immediate arm will start the intervention (telehealth visits) in Time Period 2 (following chemotherapy cycles 3 and 4). During Time Period 3 (following chemotherapy cycles 5 and 6), this arm will resume clinical care as usual.
  Interventions: Behavioral: Telehealth visits; Behavioral: Standard of Care
- Delayed Intervention Arm (Experimental): Observation periods will be from 4 days post last administration of chemotherapy until the next chemotherapy administration.
  All patients will undergo an initial observation period that will span two chemotherapy cycles and will be receiving clinical care as usual determined by the primary oncology team.
  Patients enrolled on the delayed arm will receive clinical care as usual during Time Period 2 (following chemotherapy cycles 3 and 4). During Time Period 3 (following chemotherapy cycles 5 and 6), this arm will start the intervention (telehealth visits).
  Interventions: Behavioral: Telehealth visits; Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Telehealth visits — Receiving telehealth visits with a medical provider (MD or NP) 2-3 days after last chemotherapy administration in the cycle
Behavioral: Standard of Care — Receiving care as usual from the UC Davis Comprehensive Cancer Center

SUMMARY:
This study will test the acceptability and feasibility of a telehealth intervention to improve communication between patients and medical providers in adolescent and young adult (AYA) cancer patients receiving chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer undergoing active treatment and who have received at least two cycles of chemotherapy
* Access to Epic MyChart (we will facilitate access to MyChart for interested patients who are not yet signed up)
* Access to a smartphone or tablet to access EPIC MyChart telehealth appointments

Exclusion Criteria:

* Non-English or non-Spanish speaking patients
* Potentially completing therapy during study period (including follow-up period) or plans to leave UCDCCC during study period

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients Completing the Trial | end of the study period (6 cycles of chemotherapy for each participant, where each cycle is 14-28 days)
  >65% of enrolled patients will complete the trial

SECONDARY OUTCOMES:
Survey Response Rate | end of the study period (6 cycles of chemotherapy for each participant, where each cycle is 14-28 days)
  >%70% of enrolled patients will complete the survey instruments
Telemedicine Satisfaction and Usefulness Questionnaire (TSUQ) | end of the study period (6 cycles of chemotherapy for each participant, where each cycle is 14-28 days)
  A composite score of ≥40 (based on 10 items with a Likert scale of 1-5 strongly disagree to strongly agree)

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Cancer Center, Sacramento, California, United States

REFERENCES:
- [Derived] Naz H, Apesoa-Varano EC, Romero C, Keegan T, Malogolowkin M, Callas C, Gosdin M, Alvarez E. How Do Adolescent and Young Adult Patients with Cancer Manage Their Chemotherapy-Related Symptoms at Home? J Adolesc Young Adult Oncol. 2023 Dec;12(6):923-928. doi: 10.1089/jayao.2022.0153. Epub 2023 Sep 12. PMID 37699237
- See also: Learn more or sign up for the study here! — https://studypages.com/s/improving-treatment-related-symptom-management-in-adolescents-and-young-adults-with-cancer-888566/